CLINICAL TRIAL: NCT00271453
Title: A Study to Assess the Safety, Efficacy and Pharmacokinetics of Durogesic (Fentanyl Transdermal Drug Delivery System) in the Treatment of Pediatric Patients With Chronic Pain Requiring Long-term Opioid Therapy
Brief Title: A Study to Assess the Safety and Effectiveness of Durogesic (Fentanyl Transdermal Patch) in the Treatment of Children With Chronic Pain Requiring Long-term Narcotic Pain Relief Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005950
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; opioid; fentanyl; transdermal; Durogesic; morphine
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: Durogesic® (fentanyl transdermal drug delivery system)

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of DurogesicÂ® (a transdermal patch delivering the narcotic pain-reliever fentanyl) in the treatment of children with chronic pain requiring long-term narcotic pain relief therapy.

DETAILED DESCRIPTION:
The objective of this study is to establish the analgesic efficacy, safety and pharmacokinetic profile of Durogesic® in the treatment of pediatric patients with chronic pain requiring long-term opioid therapy. Patients may be in-patients or treated at home. This study consists of three phases: a pre-trial phase, a treatment phase, and a follow-up phase. During the pre-trial phase, patients receive immediate-release oral morphine or sustained-release morphine (minimum daily dose of morphine is 30 mg/day) for at least 48 hours immediately prior to entry into the study. Patients achieving adequate pain relief in the pre-trial phase will enter the treatment phase and will be switched over to Durogesic®. The dose of Durogesic® will be calculated from the patient's daily morphine requirement, using the conversion regimen. The minimum starting dose is one patch with a fentanyl delivery rate of approximately 25 micrograms/hour. Titration in steps of 25 micrograms/hour is permitted to achieve adequate pain control. The maximum allowable dose is 300 micrograms/hour. The Durogesic® patch is applied to an area of flat skin on the upper body or upper arm, and replaced every 72 hours. The treatment phase of this study will last for 15 days (5 consecutive patch changes). Immediate-release morphine is available as rescue medication to treat breakthrough pain. Upon completion of the treatment phase, the patient may continue to receive Durogesic® therapy in the long-term follow-up phase, as long as the patient, parent or the investigator feels that it is beneficial. The primary measures of effectiveness include the patient's assessment of treatment at Day 15, pain level assessed by the patient twice daily, once in the morning and in the evening (or assessed by the parent if the patient is younger than age 5), the amount of rescue medication that the patient requires, and the pain level at the time rescue medication is given and one hour afterwards. In patients where venous access (either central or peripheral) is available, or if blood is being taken for some other purpose, blood samples will be taken to determine serum fentanyl concentrations. Safety evaluations will include the incidence of adverse events, clinical laboratory tests, assessment of the skin at the site of patch application, and vital signs. Durogesic® will be applied to the upper body or upper arm, and replaced every 72 hours. The minimum starting dose is one patch with a fentanyl delivery rate of approximately 25 micrograms/hour, titrated to achieve adequate pain control, up to a maximum dose of 300 micrograms/hour. The treatment phase is 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed malignancy (whose pain is judged by the investigator to be caused by the malignancy), or patients with other life-threatening/terminal disease whose pain requires treatment with strong opioid analgesia
* requiring treatment of pain with a strong opioid and who are expected to continue to require treatment with a strong opioid for the duration of the study
* receiving a stable dose of immediate-release oral morphine or sustained-release morphine (minimum daily dose of morphine is 30 mg/day) for at least 48 hours immediately prior to entry into the study

Exclusion Criteria:

* Patients with a history of allergy or hypersensitivity to fentanyl or morphine
* have active skin disease that precludes application of Durogesic® or which may affect the absorption of fentanyl
* have a clinical condition that in the investigator's judgment prevents participation in the study
* have participated in any other drug trial relating to pain control within one month of study entry
* currently participating in any other study or research project which would interfere with this trial.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 1996-02; Study Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Patient assessment of treatment at Day 15; Pain level assessed once in the morning and in the evening; Amount of rescue medication that the patient requires; Pain level at the time rescue medication is given and one hour afterwards

SECONDARY OUTCOMES:
Investigator and parent global assessment of the patient's treatment with respect to pain control, side effects and convenience; Pharmacokinetics; Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Hunt A, Goldman A, Devine T, Phillips M; FEN-GBR-14 Study Group. Transdermal fentanyl for pain relief in a paediatric palliative care population. Palliat Med. 2001 Sep;15(5):405-12. doi: 10.1191/026921601680419456. PMID 11591092
- See also: Click here to view the journal abstract from the study manuscript. — http://download.veritasmedicine.com/PDF/CR005824_alimentarypharmacologyandtherapeutics.pdf
- See also: A study to assess the safety and effectiveness of Durogesic� fentanyl transdermal patch in the treatment of children with chronic pain requiring long-term narcotic pain relief therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=689&filename=CR005950_CSR.pdf